CLINICAL TRIAL: NCT03734367
Title: Intervention in Emotional Intelligence in Adolescents With Type 1 Diabetes Mellitus
Brief Title: Evaluation of the Effectiveness of a Program of Emotional Intelligence in Adolescents With Type 1 Diabetes (INTEDI)
Acronym: INTEDI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Loyola Andalucia (Other)
Responsible Party: Principal Investigator, Desiree Ruiz Aranda, Doctor, Universidad Loyola Andalucia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ULoyolaAndalucia
Record Dates: First submitted 2018-10-31; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Emotional Intelligence; HbA1c; Healthy habits; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional abilities training program (Active Comparator): Intervention program on emotional abilities that will be carried out for 10 hours distributed over 5 weeks, in two and a half hour session. The work methodology will be eminently practical, working in groups including real case analysis and interactive simulation
  Interventions: Behavioral: Emotional abilities training program
- Control group (No Intervention): Control group that will not receive the training program on emotional abilities but usual care.

INTERVENTIONS:
Behavioral: Emotional abilities training program — A randomized controlled trial that evaluates the effectiveness of a program of emotional skills on metabolic control to be assessed through the glycosylated hemoglobin (HbA1c), healthy lifestyle habits and wellbeing in adolescents with type 1, Diabetes Mellitus
  Arms: Emotional abilities training program

SUMMARY:
Type 1 Diabetes Mellitus is one of the main health problems of the pediatric population worldwide, being one of the most frequent chronic endocrinology diseases in childhood and adolescence. It is a chronic degenerative disease that requires changes in the habits of life, which greatly influences the psychological functioning of those who suffer from it. Emotional factors play an important role in the control of diabetes. Specifically, emotional activation in response to different emotions such as stress, is considered one of the main factors involved in the destabilization of metabolic control in diabetes. The purpose of the study is to assess whether the introduction of a program for the development of emotional skills produces an increase in the emotional management of patients and examine whether these abilities are associated with better metabolic control measured by glycosylated hemoglobin (HbA1c), better healthy lifestyle habits and greater emotional well-being in adolescents with type 1 diabetes.This is an interventional study with two arms: 1) a control group and 2) an intervention group. The present work aims to offer a new intervention tool focused on the processing of emotional information to work the unpleasant emotions associated with this disease. The program will be designed following the Emotional Intelligence model of authors Mayer and Salovey and will focus on the development of emotional skills and knowledge that will help adolescents to promote healthy habits and improve their quality of life. The main objective of the program is to contribute to improving the knowledge and abilities of perception, assimilation, understanding and intra and interpersonal emotional regulation. The expected outcomes of the research are related to improvements in clinical practice. Increasing emotional skills of patients with diabetes can contribute to improving their quality of life and well-being. The expected results of this research will provide professionals with tools that will enable greater guarantees in adherence to treatment by patients. These results could lead to a utility model, introducing an assistance model different from the usual practice that introduces the intervention in emotional skills in the management of pediatric diabetic patients. In addition, this intervention could have an impact not only on the psychological components of the patient but also on metabolic changes and life habits.

DETAILED DESCRIPTION:
Recent research has indicated that emotional factors have an important role in the control of diabetes. According to previous literature, the burden of diabetes and its treatment contribute to emotional distress. In fact, the emotional discomfort associated with diabetes can influence the control of glycemia as it is related to the decrease of self-care behaviors and adherence to protocols and care routines. The scientific literature shows that high levels of anxiety and depression affect the adherence to treatment of diabetes, since the people who experience it are less likely to comply with health care recommendations due to the difficulty that entails compliance with the imposition of restrictions on their usual lifestyle.

The most widespread definition of emotional intelligence describes it as "the ability to accurately perceive, evaluate and express emotions; the ability to access and / or generate feelings that facilitate thinking; the ability to understand emotions and emotional knowledge; and the ability to regulate emotions promoting emotional and intellectual growth. Research shows that the ability of people to process emotional information adequately is related to effective social functioning, resilience to emotional and social pressures and less emotional impact when faced with certain health problems.

The first preliminary results of a pilot study indicated that adolescents with Type 1 Diabetes Mellitus (DM1) with high emotional abilities have a better glycemic control evaluated through HbA1c and a lower emotional discomfort associated with diabetes. These first data allow us to hypothesize that training in emotional intelligence will facilitate the increase of these skills which will contribute to the improvement of metabolic control (evaluated through HbA1c), healthy lifestyle habits and emotional well-being.

Objectives The first general objective (GO1) of our study is to design a program on emotional intelligence for intervention with adolescents with DM1 aimed at improving therapeutic adherence, healthy lifestyle habits and well-being. The second general objective (GO2) is to analyze the effectiveness of this program of improvement of emotional skills once the program is finished, 6 and 12 months after the intervention.

Pre-intervention phase: The specific objectives (SO) are:

* (SO1) Development of the intervention sessions and preparation of theoretical materials and practical dynamics.
* (SO2) Evaluate the adequacy of the contents and methodology of the program through a focus group and individualized interviews with the target population.

(OG2) Analyze the effectiveness of this program to improve emotional skills once the program ends, at 6 and 12 months after the intervention.

Intervention Phase: The specific objectives (SO) are:

* (SO3) Evaluate the psychological and metabolic variables of adolescents with DM1 prior to the intervention of the control group and the intervention group to establish the baseline.
* (SO4) Implementation of the intervention program in the intervention group during 5 sessions of 2 and a half hours.
* (SO5) Evaluate the psychological and metabolic variables of adolescents with DM1 in the control group and in the intervention group after the end of the program.

Follow-up phase: The specific objectives (SO) are

-(SO6) To evaluate the psychological and metabolic variables of adolescents with DM1 in the control group and intervention group at 6 and 12 months after the program to analyze the maintenance of the results.

Methods Participants Participants will be recruited from a University Hospital Virgen Macarena. The estimation for the sample size is based on the average HbA1c of 8.84% (±1.39) (73.1± 15.3 mmol/mol) in adolescents between 11 and 16 years of age (n = 133) with a diagnosis of less than one year indicating that 31 participants will be needed per group to achieve an 80% probability of detecting a difference of 1% (11 mmol/mol) in HbA1c means between the two groups with a significance of 5%. It will be emphasized that participation in the study is voluntary. Participants may withdraw from it in any moment.

Procedure

According to the objectives set, the research project is structured in different phases:

A) PRE-INTERVENTION PHASE:

1. Development of the intervention sessions and preparation of theoretical and dynamic materials practices. The adequacy of the contents and methodology of the program will be evaluated through of a focus group and individualized interviews with the target population.
2. Adolescents will be recruited through specialist physicians in the area of University Hospital Virgen Macarena. The participants and their parents / guardians will be informed by the principal investigator of the nature of the study, its usefulness, the mode of realization and the people involved.
3. Consent and informed consent will be administered by the investigator principal along with a fact sheet on the objectives and procedure of the investigation as well as the data of the project contact person.
4. Participants will be assigned randomly to each of the groups. For it a simple random assignment will be made using the procedure "Assignment of subject to treatments "available in 'Epidat software' version 3.1.
5. The following data will be collected: Sociodemographic variables, clinical variables, metabolic control variables, psychological variables

   B) INTERVENTION PHASE
6. A program of intervention in emotional skills will be carried out. The work methodology will be eminently practical, working in groups including analysis of real cases and interactive simulation.
7. After the intervention, the psychological team will carry out the evaluation of the variables, as well as the collection of clinical, biochemical, of metabolic control, healthy living habits and emotional well-being.
8. Parents of adolescents will receive two training sessions in emotional skills of two hour each with the objective of helping adolescents to consolidate the contents and skills acquired during the intervention program.

   C) FOLLOW-UP PHASE
9. In the third year of the project, 2 sessions will be held to know if participants had any problems with what they learned in the intervention, remember the principles and main techniques for its implementation.
10. At months 6 and 12 after the intervention, there will be a re-evaluation of psychological and metabolic control variables to analyze the maintenance of the results.
11. If the intervention achieves the proposed objectives, once the study is completed, the adolescents of the control group will be offered to participate in the intervention program.

Design This is a randomized controlled trial that evaluates the effectiveness of a program of emotional skills on metabolic control, healthy lifestyle habits and well-being with two groups (intervention group and control group) with pre-post-treatment measures and follow-up.

Materials

* Perceived emotional intelligence (TMMS-24)
* Scale of positive and negative affect (PANAS)
* Difficulties in Emotion Regulation Scale (DERS)
* Diabetes-related Distress Scale (DDS-17)
* Diet and Exercise domain of the (eVITAL Toolkit)
* Health questionnaire (SF-36)

Analysis of data The results will be analyzed according to the objectives proposed in the project. The effectiveness of the intervention in the increase of the emotional skills and the improvement of the metabolic control, healthy habits and emotional well-being will be estimated comparing the pre and post evaluations of the group intervention through different statistics of comparison of means such as the non-parametric Wilcoxon statistic and the pre-post-follow-up measures with the nonparametric statistic for repeated Friedman measurements. ANCOVA analysis of covariance will be used in order to separate the effect of the intervention from the effect of the differences in the selection of the participants. To check the effectiveness of the intervention, analysis of the covariance on the post-test will be carried out for both groups (intervention and control) including as a covariate the scores in the pre-test.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of type 1 Diabetes Mellitus for at least 12 months.
* Type of treatment, International Unit insulin/kg

Exclusion Criteria:

* Present some incapacitating psychiatric disorder or other chronic illness.
* Not giving informed consent

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in emotional skills of adolescents with type 1 diabetes related to a greater emotional regulation | Pre-test (before intervention), post-test (after the intervention; month 6 and month 12)
  Participants will be asked to complete a battery of psychological questionnaires
  -Difficulties in Emotion Regulation Scale (DERS) This is a 28-item, self-report questionnaire measuring clinically relevant difficulties in emotion regulation. In the Spanish adaptation, the items are grouped into five subscales: impulse control difficulties, non-acceptance of emotional response, difficulties engaging in goal-directed behavior, lack of emotional awareness and lack of emotional clarity. Subscales are scored on a 5-point scale ranging from 1 (never) to 5 (always). Higher scores indicate greater difficulty with emotion regulation. This scale has been shown to have adequate psychometric properties.
Change in emotional skills of adolescents with type 1 diabetes related to less stress levels | Pre-test (before intervention), post-test (after the intervention; month 6 and month 12)
  Participants will be asked to complete a battery of psychological questionnaires
  -The Diabetes Distress Scale (DDS-17). It assesses the emotional distress associated with diabetes and it includes four dimensions: emotional burden, physician-related distress, regimen-related distress, and diabetes-related interpersonal distress. Higher scores indicate greater stress related to disease. This scale has been shown to have adequate internal consistency and validity. Cronbach's alpha ranged from 0.88 to 0.93
Change in emotional skills of adolescents with type 1 diabetes related to a greater positive affect | Pre-test (before intervention), post-test (after the intervention; month 6 and month 12)
  Participants will be asked to complete a battery of psychological questionnaires
  -Positive and Negative Affect Schedule (PANAS). It is a self-reported adjective checklist that contains two 20-item subscales designed for the assessment of positive and negative affect. Respondents use a 5-point Likert scale to rate the extent to which they usually feel each of 20 emotion-related words. Reliability and validity reported by Watson and colleagues was moderately good. Cronbach's alpha ranged from 0.87 to 0.90.
Change in emotional skills of adolescents with type 1 diabetes related to an increase in healthy life habits | Pre-test (before intervention), post-test (after the intervention; month 6 and month 12)
  Participants will be asked to complete a battery of psychological questionnaires
  -eVITAL toolkit8. Adaptation of the Macrodomain Diet and Exercise 4.1 Domain diet and nutrition and 4.2. Domain exercise eVITAL toolkit for measuring healthy habits in diabetes.
Change in emotional skills of adolescents with type 1 diabetes related to a greater perception of quality of life | Pre-test (before intervention), post-test (after the intervention; month 6 and month 12)
  Participants will be asked to complete a battery of psychological questionnaires
  -The PedsQL 4.0 Generic Core Scales. The 23-item PedsQL 4.0 Generic Core Scales comprise four multi-item scales that explore dimensions of health-related quality of life: 1) physical functioning (8 items), 2) emotional functioning (5 items), 3) social functioning (5 items), and 4) school functioning (5 items). Respondents use a 5-point Likert scale. Higher scores indicate greater quality of life.
Change in the emotional skills of adolescents with type 1 diabetes that will be related to a glycosylated index between normal values | Pre-test (before intervention), post-test (after the intervention; month 6 and month 12)
  Metabolic variables will be assessed using a flash glucose monitoring (FGM) device.
  Glycemic control. Participants report their HbA1c level from their last blood test. The American Diabetes Association recommends a target HbA1c of 7.5% for children and adolescents. Moreover, mean glucose, standard deviation, percentage of glucose in normoglycemia (time in range, according to individualized target), percent of time in hypoglycemia (below 70) and percent of time in hyperglycemia (according to an individualized target), and number of hypoglycemic episodes will be collected. Variables will be analyzed from the last 15 days prior to evaluation. Metabolic variables will be obtained using a flash glucose monitoring (FMG) device (Free Style Libre) as it has become the standard glucose monitoring system in the Andalusian Public Health System for the pediatric population. For non-FMG users, metabolic variables will be obtained by glucometers through their specific software.

CONTACTS AND LOCATIONS:
Overall Officials: Desireé Ruiz, Psychologist, Principal Investigator — Universidad Loyola Andalucía
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ruiz-Aranda D, Extremera N, Pineda-Galan C. Emotional intelligence, life satisfaction and subjective happiness in female student health professionals: the mediating effect of perceived stress. J Psychiatr Ment Health Nurs. 2014 Mar;21(2):106-13. doi: 10.1111/jpm.12052. Epub 2013 Apr 12. PMID 23578272
- [Background] Ruiz-Aranda D, Salguero JM, Fernandez-Berrocal P. Emotional intelligence and acute pain: the mediating effect of negative affect. J Pain. 2011 Nov;12(11):1190-6. doi: 10.1016/j.jpain.2011.06.008. Epub 2011 Aug 23. PMID 21865092
- [Result] Ruiz-Aranda D, Zysberg L, Garcia-Linares E, Castellano-Guerrero AM, Martinez-Brocca MA, Gutierrez-Colosia MR. Emotional abilities and HbA1c levels in patients with type 1 diabetes. Psychoneuroendocrinology. 2018 Jul;93:118-123. doi: 10.1016/j.psyneuen.2018.04.015. Epub 2018 Apr 20. PMID 29723781
- [Derived] Ruiz-Aranda D, Resurreccion DM, Gutierrez-Colosia MR, Martinez-Brocca MA. Intervention in emotional abilities for adolescents with type 1 diabetes mellitus in a hospital setting: a study protocol for a randomised controlled trial. BMJ Open. 2019 Aug 27;9(8):e027913. doi: 10.1136/bmjopen-2018-027913. PMID 31462466